CLINICAL TRIAL: NCT01134952
Title: A Prospective Cross-over Study Comparing the Effect of Sirolimus Versus Mycophenolate on Viral Load in Liver Transplant Recipients With Recurrent Chronic HCV Infection
Brief Title: Study of Sirolimus Versus Mycophenolate Liver Transplant Recipients With Recurrent Hepatitis C Virus (HCV)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Vivian McAlister, Principal investigator, London Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UWO12961
Record Dates: First submitted 2010-05-27; First posted 2010-06-02 (Estimated); Results first posted 2015-01-21 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Hepatitis C
Keywords: sirolimus; everolimus; mycophenolic acid; hepatitis C virus; tacrolimus; viral load
MeSH Terms: conditions — Hepatitis C | interventions — Sirolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mycophenolate to sirolimus switch (Experimental): Liver transplant recipients with Hepatitis C virus switched from mycophenolate mofetil (MMF) to sirolimus (SRL) for 3 months and then switched back to MMF
  Interventions: Drug: Mycophenolate to sirolimus switch

INTERVENTIONS:
Drug: Mycophenolate to sirolimus switch — Sirolimus given for 3 months instead of mycophenolate at a starting dose equivalent of 1 mg sirolimus equal to 1000 mg of mycophenolate.
  Other Names: rapamune; rapamycin; mycophenolic mofetil; mycophenolic acid; cellcept

SUMMARY:
Different immunosuppressive drugs used in transplantation may reduce the body's defences against infection differently. It is known that patients with Hepatitis C virus, known as HCV, who switched from azathioprine to mycophenolate mofetil experienced an increase in viral load. Despite this, mycophenolate mofetil is used because it prevents rejection more reliably than azathioprine. Sirolimus is an another immunosuppressive agent that reliably prevents rejection and may have antiviral activity. This study is designed to see if the viral load of HCV and other viruses is reduced by switching from mycophenolate to sirolimus.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) persistence after liver transplantation for HCV end-stage liver disease is universal and in this clinical setting, HCV mediated liver injury has been reported to follow a more progressive course compared to the non-immunosuppressed patient. Additionally, patients with recurrent chronic hepatitis C develop higher viral load compared to pre-transplant levels. Such persistently high viral burden post transplant may contribute to allograft damage. The choice of calcineurin inhibitor (CNI) does not effect recurrence rates of HCV hepatitis. HCV is also associated with renal dysfunction so that reduction in exposure to calcineurin inhibitors (CNI) is desirable. Unfortunately steroids are associated with a marked increase in HCV replication and cannot be used to reduce CNI doses. Mycophenolate mofetil (MMF) increases HCV viral load. A recent increase in the severity of recurrent hepatitis in patients with HCV receiving liver transplants has been attributed to MMF and interleukin-2 receptor blockers. Increased fibrosis of the liver occurs during antiviral anti HCV treatment in patients taking mycophenolate but patients on azathioprine develop cirrhosis faster, possibly because of rejection.

A large industry sponsored phase III clinical trial has been underway for several years where patients have substituted sirolimus (SRL) for calcineurin inhibitors after liver transplantation. The object of that study is to determine impact of conversion on renal function. No detrimental effect (thrombosis, rejection or recurrent viral infection) was apparent to the safety board after two reviews. No study has compared SRL to MMF after liver transplantation.

SRL, an immunosuppressive drug that inhibits the activation and proliferation of T-lymphocytes, is associated with reduction of Epstein Barr Virus (EBV) post-transplantation viral load in children. Experimentally it inhibits the growth of EBV B-cell lymphoma. A pilot study of tacrolimus with SRL showed a powerful anti-rejection effect but a subsequent trial was halted early because of an increase in hepatic artery thrombosis even though the rates of thrombosis in either arm of the study was below that expected. A recent large series in patients with hepatocellular carcinoma (most of whom had HCV) who received large doses of SRL showed a beneficial anti-cancer effect without thrombosis. The randomised trials and the reported series all had large numbers of patients with HCV. The absence of obvious recurrent HCV hepatitis and the low rates of cytomegalovirus (CMV) disease coupled with the known inhibition of EBV replication gives hope that SRL has anti-viral properties at immunosuppressive doses. Early reports confirm that hope: 1) successful liver transplantation in patients with HIV and HCV. "Significantly better control of HIV and HCV replication was found among patients taking RAPA monotherapy (P=0.0001 and 0.03, respectively)"; 2) switching to sirolimus in renal transplant recipients with hepatitis C virus: HCV replication reduced by switch to sirolimus; 3) sustained, spontaneous disappearance of serum HCV-RNA under immunosuppression after liver transplantation for HCV cirrhosis: two liver recipients who spontaneously cleared HCV after switch to sirolimus.

SRL (2 mg/day) and MMF (2g/day) are licensed as adjuvant immunosuppressive agents to be used in kidney transplantation with cyclosporine so that immunosuppressive equivalent doses are 1mg SRL = 1g MMF.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent HCV after liver transplantation
* Taking mycophenolate mofetil
* Stable liver function

Exclusion Criteria:

* Pregnant females or couples unwilling to use contraception
* Intolerance or allergy to sirolimus
* Patients taking anti-HCV therapy
* Patients taking medications known to alter the levels of sirolimus
* History of thromboembolic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivian McAlister, MB, FRCSC, Study Director — London Health Sciences Centre; Natasha Chandok, MD, FRCPC, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Background] Zekry A, Gleeson M, Guney S, McCaughan GW. A prospective cross-over study comparing the effect of mycophenolate versus azathioprine on allograft function and viral load in liver transplant recipients with recurrent chronic HCV infection. Liver Transpl. 2004 Jan;10(1):52-7. doi: 10.1002/lt.20000. PMID 14755778
- [Background] McAlister VC, Gao Z, Peltekian K, Domingues J, Mahalati K, MacDonald AS. Sirolimus-tacrolimus combination immunosuppression. Lancet. 2000 Jan 29;355(9201):376-7. doi: 10.1016/S0140-6736(99)03882-9. PMID 10665560
- [Background] Di Benedetto F, Di Sandro S, De Ruvo N, Montalti R, Ballarin R, Guerrini GP, Spaggiari M, Guaraldi G, Gerunda G. First report on a series of HIV patients undergoing rapamycin monotherapy after liver transplantation. Transplantation. 2010 Mar 27;89(6):733-8. doi: 10.1097/TP.0b013e3181c7dcc0. PMID 20048692
- [Background] Gallego R, Henriquez F, Oliva E, Camacho R, Hernandez R, Hortal L, Sablon N, Quintana B, Santana R, Gonzalez F, Palop L, Vega N. Switching to sirolimus in renal transplant recipients with hepatitis C virus: a safe option. Transplant Proc. 2009 Jul-Aug;41(6):2334-6. doi: 10.1016/j.transproceed.2009.06.064. PMID 19715912
- [Background] Samonakis DN, Cholongitas E, Triantos CK, Griffiths P, Dhillon AP, Thalheimer U, Patch DW, Burroughs AK. Sustained, spontaneous disappearance of serum HCV-RNA under immunosuppression after liver transplantation for HCV cirrhosis. J Hepatol. 2005 Dec;43(6):1091-3. doi: 10.1016/j.jhep.2005.08.005. Epub 2005 Sep 15. PMID 16239045
- [Background] Ballardini G, De Raffele E, Groff P, Bioulac-Sage P, Grassi A, Ghetti S, Susca M, Strazzabosco M, Bellusci R, Iemmolo RM, Grazi G, Zauli D, Cavallari A, Bianchi FB. Timing of reinfection and mechanisms of hepatocellular damage in transplanted hepatitis C virus-reinfected liver. Liver Transpl. 2002 Jan;8(1):10-20. doi: 10.1053/jlts.2002.30141. PMID 11799480
- [Background] Charlton M. Liver biopsy, viral kinetics, and the impact of viremia on severity of hepatitis C virus recurrence. Liver Transpl. 2003 Nov;9(11):S58-62. doi: 10.1053/jlts.2003.50245. PMID 14586897
- [Background] Sindhi R, Webber S, Venkataramanan R, McGhee W, Phillips S, Smith A, Baird C, Iurlano K, Mazariegos G, Cooperstone B, Holt DW, Zeevi A, Fung JJ, Reyes J. Sirolimus for rescue and primary immunosuppression in transplanted children receiving tacrolimus. Transplantation. 2001 Sep 15;72(5):851-5. doi: 10.1097/00007890-200109150-00019. PMID 11571449
- [Background] Nepomuceno RR, Balatoni CE, Natkunam Y, Snow AL, Krams SM, Martinez OM. Rapamycin inhibits the interleukin 10 signal transduction pathway and the growth of Epstein Barr virus B-cell lymphomas. Cancer Res. 2003 Aug 1;63(15):4472-80. PMID 12907620
- [Background] Kneteman NM, Oberholzer J, Al Saghier M, Meeberg GA, Blitz M, Ma MM, Wong WW, Gutfreund K, Mason AL, Jewell LD, Shapiro AM, Bain VG, Bigam DL. Sirolimus-based immunosuppression for liver transplantation in the presence of extended criteria for hepatocellular carcinoma. Liver Transpl. 2004 Oct;10(10):1301-11. doi: 10.1002/lt.20237. PMID 15376305
- [Background] Iacob S, Cicinnati VR, Hilgard P, Iacob RA, Gheorghe LS, Popescu I, Frilling A, Malago M, Gerken G, Broelsch CE, Beckebaum S. Predictors of graft and patient survival in hepatitis C virus (HCV) recipients: model to predict HCV cirrhosis after liver transplantation. Transplantation. 2007 Jul 15;84(1):56-63. doi: 10.1097/01.tp.0000267916.36343.ca. PMID 17627238
- [Background] Kornberg A, Kupper B, Tannapfel A, Hommann M, Scheele J. Impact of mycophenolate mofetil versus azathioprine on early recurrence of hepatitis C after liver transplantation. Int Immunopharmacol. 2005 Jan;5(1):107-15. doi: 10.1016/j.intimp.2004.09.010. PMID 15589468
- [Background] Haddad EM, McAlister VC, Renouf E, Malthaner R, Kjaer MS, Gluud LL. Cyclosporin versus tacrolimus for liver transplanted patients. Cochrane Database Syst Rev. 2006 Oct 18;2006(4):CD005161. doi: 10.1002/14651858.CD005161.pub2. PMID 17054241
- [Background] Rostaing L, Izopet J, Sandres K, Cisterne JM, Puel J, Durand D. Changes in hepatitis C virus RNA viremia concentrations in long-term renal transplant patients after introduction of mycophenolate mofetil. Transplantation. 2000 Mar 15;69(5):991-4. doi: 10.1097/00007890-200003150-00055. PMID 10755563
- See also: Transplant Program website — http://www.lhsc.on.ca/About_Us/MOTP/

RESULTS

PARTICIPANT FLOW:
Groups:
- MMF SRL Switch: Liver transplant recipients with Hepatitis C virus taking sirolimus (SRL) instead of mycophenolate mofetil (MMF) for 3 months
Period: Overall Study
Arm/Group | MMF SRL Switch
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- MMF MRL Switch: Liver transplant recipients with Hepatitis C virus switched from mycophenolate mofetil (MMF) to sirolimus (SRL) for 3 months and then switched back to MMF
Arm/Group | MMF MRL Switch
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 8
Region of Enrollment [Number; unit: participants]
  Canada | 11
Hepatitis C viral load [Mean (Standard Deviation); unit: 10^7 HCV IU/mL] | 2.8 (2.6)
Tacrolimus trough level [Mean (Standard Deviation); unit: ng/ml] | 5.5 (1.9)
Bilirubin [Mean (Standard Deviation); unit: umol/L] | 8.8 (3.2)
Alkaline phosphatase [Mean (Standard Deviation); unit: U/L] | 94.5 (40.2)
Alanine aminotransferase [Mean (Standard Deviation); unit: U/ml] | 86.3 (56.1)
Hemoglobin [Mean (Standard Deviation); unit: g/L] | 145.1 (13.2)
Platelet count [Mean (Standard Deviation); unit: 10^9/L] | 165.3 (58.3)
Fasting cholesterol [Mean (Standard Deviation); unit: mmol/L] | 4.9 (1.4)
Triglyceride [Mean (Standard Deviation); unit: mmol/L] | 1.7 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Delta Hepatitis C Viral Load
Description: Percent change in HCV load determined 3 months after switch from MMF to SRL.
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- MMF SRL Switch: Liver transplant recipients with HCV 3 months after switch from mycophenolate to sirolimus
Arm/Group | MMF SRL Switch
Number analyzed (Participants) | 11
percent change | 15 (53)

2. Secondary Outcome: Final Hepatitis C Viral Load
Description: Percent change in HCV load determined 3 months after switch from SRL to MMF
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- MMF SRL Switch: All patients switched for 3 months from mycophenolate mofetil to sirolimus and then back to mycophenolate mofetil
Arm/Group | MMF SRL Switch
Number analyzed (Participants) | 11
percent change | -47 (100)

3. Secondary Outcome: Sirolimus Trough Level
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- MMF SRL Switch: All patients after switch from mycophenolate to sirolimus
Arm/Group | MMF SRL Switch
Number analyzed (Participants) | 11
ng/ml | 7.2 (2.2)

4. Secondary Outcome: Delta Tacrolimus Trough Level
Description: Percent change determined 3 months after switch from MMF to SRL
Time Frame: 3 month
Population: 2 patients did not have tacrolimus levels recorded during both time periods and are excluded
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- MMF SRL Switch: Liver transplant recipients switched from mycophenolate mofetil to sirolimus
Arm/Group | MMF SRL Switch
Number analyzed (Participants) | 9
percent change | 23 (82)

5. Secondary Outcome: Delta Bilirubin
Description: Percent change determined 3 months after switch from MMF to SRL
Time Frame: 3 month
Population: Levels available at correct time in only 7 patients
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- MMF SRL Switch: All patients 3 months after switch from mycophenolate to sirolimus
Arm/Group | MMF SRL Switch
Number analyzed (Participants) | 7
percent change | -6.0 (25)

6. Secondary Outcome: Delta Alkaline Phosphatase
Description: Percent change determined 3 months after switch from MMF to SRL
Time Frame: 3 month
Population: Levels not available at appropriate times in 2 patients
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | MMF SRL Switch
Number analyzed (Participants) | 9
percent change | 13.8 (3)

7. Secondary Outcome: Delta Alanine Aminotransferase
Description: Percent change determined 3 months after switch from MMF to SRL
Time Frame: 3 month
Population: Levels at appropriate time not available in 2 patients
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | MMF SRL Switch
Number analyzed (Participants) | 9
percent change | 9 (28)

8. Secondary Outcome: Delta Hemoglobin
Description: Percent change determined 3 months after switch from MMF to SRL
Time Frame: 3 month
Population: Levels at appropriate times not available in 2 patients
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | MMF SRL Switch
Number analyzed (Participants) | 9
percent change | -2.7 (2.7)

9. Secondary Outcome: Delta Platelet Count
Description: Percent change determined 3 months after switch from MMF to SRL
Time Frame: 3 month
Population: Levels not available on 2 patients at appropriate time
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | MMF SRL Switch
Number analyzed (Participants) | 9
percent change | -8.5 (20)

10. Secondary Outcome: Delta Cholesterol Fasting Level
Description: Percent change determined 3 months after switch from MMF to SRL
Time Frame: 3 month
Population: Levels not available for 2 patients
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | MMF SRL Switch
Number analyzed (Participants) | 9
percent change | 1.2 (55)

11. Secondary Outcome: Delta Triglyceride Fasting Level
Description: Percent change determined 3 months after switch from MMF to SRL
Time Frame: 3 month
Population: Levels at appropriate times not available on 2 patients
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | MMF SRL Switch
Number analyzed (Participants) | 9
percent change | 23 (81)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- MMF SRL Switch: All patients during 3 month period of switch from mycophenolate mofetil (MMF) to sirolimus and for 3 months after switch back to MMF
Arm/Group | MMF SRL Switch
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

LIMITATIONS AND CAVEATS:
Greater than expected baseline variation; technical problems with laboratory measurement of HCV (two different platforms used); and poor recruitment over a long period make the results difficult to interpret.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No